CLINICAL TRIAL: NCT02378883
Title: Apollo™ Onyx™ Delivery Microcatheter Post Market Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV-APL001
Record Dates: First submitted 2015-02-24; First posted 2015-03-04 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-03

CONDITIONS: Arteriovenous Malformations
Keywords: Apollo; Onyx; Arteriovenous malformation; AVM; Onyx™ Liquid Embolic System; Apollo™ Onyx™ Delivery Microcatheter; Brain Diseases
MeSH Terms: conditions — Arteriovenous Malformations; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVM treatment (Other): Apollo™ Onyx™ Delivery Micro Catheter
  Interventions: Device: Apollo™ Onyx™ Delivery Micro Catheter

INTERVENTIONS:
Device: Apollo™ Onyx™ Delivery Micro Catheter

SUMMARY:
The purpose of this study is to evaluate the safety of the Apollo™ Onyx™ Delivery Microcatheter used for delivery of the Onyx™ Liquid Embolic System during brain arteriovenous malformation (AVM) embolization procedures.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, multicenter, post-market safety evaluation of subjects indicated for embolization of brain AVMs with the study device. The study device was developed to potentially minimize the side effects of catheter retainment and increased procedural risk associated with alternative methods necessary for removing entrapped catheters. In the event of catheter retainment, using the Apollo™ Onyx™ Delivery Microcatheter versus any a standard catheter represents leaving behind a 1.5 - 3.0 cm long detachable tip in the Onyx™ Onyx™ Delivery Microcatheter cast versus an average 165 cm long catheter in the vasculature.

ELIGIBILITY:
Inclusion Criteria:

* The Subject or Subject's legally authorized representative has signed and dated an informed consent form.
* The Subject has a confirmed diagnosis of a brain AVM.
* The Subject is clinically and neurologically stable for a minimum of 48 hours prior to embolization.
* The Subject has a life expectancy of at least 1 year.
* The Subject agrees to and is capable of completing all study-required procedures.

Exclusion Criteria:

* Current participation in another investigational drug or device study that evaluates treatments for brain AVMs or other cerebrovascular disease.
* The Subject has a bleeding disorder.
* The Subject is not a candidate for the use of vasodilators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Aziz-Sultan, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Radiology Imaging Associates, P.C., Englewood, Colorado
  - Brigham's & Women Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Generally we do not plan to share the IPD. Researchers can contact the Sponsor if interested.

REFERENCES:
- [Derived] Meyers PM, Fifi JT, Cockroft KM, Miller TR, Given CA, Zomorodi AR, Jagadeesan BD, Mokin M, Kan P, Yao TL, Diaz O, Huddle D, Bellon RJ, Seinfeld J, Polifka AJ, Fiorella D, Chitale RV, Kvamme P, Morrow JT, Singer J, Wakhloo AK, Puri AS, Deshmukh VR, Hanel RA, Gonzalez LF, Woo HH, Aziz-Sultan MA. Safety of the APOLLO Onyx delivery microcatheter for embolization of brain arteriovenous malformations: results from a prospective post-market study. J Neurointerv Surg. 2021 Oct;13(10):935-941. doi: 10.1136/neurintsurg-2020-016830. Epub 2021 Feb 1. PMID 33526480

RESULTS

PARTICIPANT FLOW:
Groups:
- APOLLO: The Apollo™ Onyx™ Delivery Microcatheter used for delivery of the Onyx™ Liquid Embolic System during brain AVM embolization procedures.
Period: Enrollment
Arm/Group | APOLLO
Started | 121 (Participants consented and assessed for eligibility)
Completed | 112 (Attempted with study device - intent to treat population)
Not Completed | 9
Not completed — Subject did not meet Inclusion criteria | 6
Not completed — Attempt to use Apollo was not performed | 3
Period: Discharge
Arm/Group | APOLLO
Started | 112
Completed | 112
Not Completed | 0
Period: 30 Day Follow-Up
Arm/Group | APOLLO
Started | 112
Completed (Includes 66 subjects with no tip retained. Subjects eligible to exit study per protocol.) | 106
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2
Not completed — Missed Visit | 2
Not completed — Death | 1
Period: 12 Months Follow-Up
Arm/Group | APOLLO
Started (As per protocol only 46 subjects were eligible for 12 month visit due to tip retention.) | 46 (Two deaths occurred between 30 day FU and prior to 12 month FU.)
Completed | 41
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | APOLLO
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 90
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 79
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  United States | 112
Smoking [Count of Participants; unit: Participants]
  Never smoked or not smoked within last 10 yrs | 54
  Not a current smoker but has smoked in past 10 yrs | 23
  Current smoker, less than one pack per day | 19
  Current smoker more than or equal to one pack/day | 13
  Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Catheter-related Adverse Events at 30 Days
Description: Premature (unintentional) catheter tip detachment with clinical sequelae
  Catheter rupture/break/fracture with clinical sequelae
  Retained catheter body in the vasculature
Time Frame: 30 days, after treatment with Onyx™ embolization using Apollo™ Onyx™ Delivery Microcatheter
Population: The Apollo™ Onyx™ Delivery Microcatheter used for delivery of the Onyx™ Liquid Embolic System during brain AVM embolization procedures.
Measure: Count of Participants; unit: Participants
Groups:
- AVM Treatment: Apollo™ Onyx™ Delivery Microcatheter
Arm/Group | AVM Treatment
Number analyzed (Participants) | 112
Participants | 0

2. Secondary Outcome: Number of Participants With Premature (Unintentional) Catheter Tip Detachment at 30 Days
Description: Rate of premature (unintentional) catheter tip detachment
Time Frame: 30 days
Population: Participants treated with Onyx™ embolization using Apollo™ Onyx™ Delivery Microcatheter
Measure: Count of Participants; unit: Participants
Arm/Group | APOLLO
Number analyzed (Participants) | 112
Participants | 1

3. Secondary Outcome: Number of Participants With Intentional Catheter Tip Detachment at 30 Days
Description: Rate of intentional catheter tip detachment
Time Frame: 30 days
Population: Participants treated with Onyx™ embolization using Apollo™ Onyx™ Delivery Microcatheter
Measure: Count of Participants; unit: Participants
Arm/Group | APOLLO
Number analyzed (Participants) | 112
Participants | 68

4. Secondary Outcome: Number of Participants With Migration of Retained Catheter Tip Post Embolization at 30 Days
Description: Rate of migration of the retained catheter tip post embolization
Time Frame: 30 days
Population: Participants treated with Onyx™ embolization using Apollo™ Onyx™ Delivery Microcatheter
Measure: Count of Participants; unit: Participants
Arm/Group | APOLLO
Number analyzed (Participants) | 112
Participants | 0

5. Secondary Outcome: Number of Participants With Catheter/Tip Leakage From Detachment Zone at 30 Days
Description: Rate of catheter/tip leakage from detachment zone
Time Frame: 30 days
Population: Participants treated with Onyx™ embolization using Apollo™ Onyx™ Delivery Microcatheter
Measure: Count of Participants; unit: Participants
Arm/Group | APOLLO
Number analyzed (Participants) | 112
Participants | 0

6. Secondary Outcome: Number of Participants With Catheter-related Adverse Events at 30 Days
Description: Incidence of catheter-related adverse events at 30 days
Time Frame: 30 days
Population: Participants treated with Onyx™ embolization using Apollo™ Onyx™ Delivery Microcatheter
Measure: Count of Participants; unit: Participants
Arm/Group | APOLLO
Number analyzed (Participants) | 112
Participants | 31

7. Secondary Outcome: Number of Participants With Catheter-related Adverse Events at 12 Months
Description: Number of participants with catheter-related adverse events at 12 months (long term secondary endpoint)
Time Frame: 12 months
Population: Participants treated with Onyx™ embolization using Apollo™ Onyx™ Delivery Microcatheter
Measure: Count of Participants; unit: Participants
Arm/Group | APOLLO
Number analyzed (Participants) | 112
Participants | 68

8. Secondary Outcome: Number of Participants With Migration of Retained Catheter Tip Post Embolization at 12 Months
Description: Rate of migration of the retained catheter tip post embolization (long-term secondary endpoint)
Time Frame: 12 months
Population: Participants treated with Onyx™ embolization using Apollo™ Onyx™ Delivery Microcatheter
Measure: Count of Participants; unit: Participants
Arm/Group | APOLLO
Number analyzed (Participants) | 112
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the point of enrollment in the study until a subject exited the study (at 30-days or 12-months)
Description: The adverse event data was adjudicated by a three member independent Clinical Events Committee (CEC). All data presented within this section has been CEC adjudicated. Adjudicable events met the following criteria:
  * All Serious Adverse Events (SAEs)
  * All device-related Adverse Events
  * All procedure-related Adverse Events
  * All AEs with an underlying neurological cause (neurological adverse event)
Arm/Group | APOLLO
All-Cause Mortality (participants affected / at risk) | 3/112
Serious Adverse Events (participants affected / at risk) | 39/112
Other Adverse Events (participants affected / at risk) | 51/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APOLLO (N=112)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 4 (4)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Hemianopia (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 6 (6)
Migraine (Nervous system disorders) | 1 (1)
Monoparesis (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Air embolism (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Vessel perforation (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APOLLO (N=112)
Bradycardia (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 4 (4)
Photophobia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 4 (4)
Visual impairment (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Adverse drug reaction (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Pneumocephalus (Injury, poisoning and procedural complications) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 2 (2)
Cerebral artery thrombosis (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebral vasoconstriction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysmetria (Nervous system disorders) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 17 (18)
Hemianopia homonymous (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2)
Quadrantanopia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 8 (9)
Vertebral artery dissection (Nervous system disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 8 (11)

LIMITATIONS AND CAVEATS:
Study was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT02378883/Prot_SAP_000.pdf